CLINICAL TRIAL: NCT03007108
Title: Determination of Normal Range Values of Thrombin Generation Parameters in Pediatrics Population Using a New Standardized Thrombin Generation Assay
Brief Title: Age-dependency of Thrombin Generation Using a New Standardized Assay
Acronym: TGT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PO16107
Record Dates: First submitted 2016-12-27; First posted 2017-01-02 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Healthy Infants

ARMS (1):
- healthy infants (Experimental)
  Interventions: Other: blood withdrawal

INTERVENTIONS:
Other: blood withdrawal

SUMMARY:
The aim of this study is to establish normal values of thrombin generation assay parameters in pediatrics, according to different age groups. The standardized thrombin generation assay "Genesia™" will be used. Different age groups of healthy children will be recruited : neonates, 1-3 months, 3-6 months, 6-12 months, 1-2 years, 2-6 years, 6-12 years, and 12-15 years old. Adults values will be obtained (healthy adults > 18 years old).

DETAILED DESCRIPTION:
Materials and Methods Collection of blood samples Blood samples of 240 healthy children will be obtained from the blood that will be collected for the routine coagulation screening (in neonates and in children < 18 months) or at the time of surgery in children aged > 18 months. Healthy neonates will be recruited by the neonatologists. Children aged from 1 month to 15 years will be included by anesthesiologists before minor elective surgery such as tonsillectomy, adenoidectomy, phimosis or oral surgery. Additionally, blood from adults referred for thrombophilia testing will be studied. This study was approved by French authorities (ANSM and CPP). Inform consent will be obtained from all participants. Blood will be collected into plastic tubes containing sodium citrate (0.106 M, tubes from "Starstedt"). Platelet poor plasma will be obtained by two centrifugations for 10 minutes at 2500 g at room temperature and stored at - 70°C until further examination.

Statistical analysis Statistical analysis will be performed as 1) a descriptive analysis (frequency and percentage for qualitative data, mean, SD and centiles for quantitative data), and 2) a comparison analysis (student, Mann-Withney, Kruskall- Wallis).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent from parents of children
* Informed consent from patients in the case of adults refered for thrombophilia testing
* Affiliation to the French Health Social System

Exclusion Criteria:

* weight < 3250 g
* Patients under law protection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Thrombin generation | Day 0
  The standardized thrombin generation assay Genesia™ will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France